CLINICAL TRIAL: NCT02919488
Title: The Effect of an Acute Bout of Exercise on High-sugar Meal Induced Endothelial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Meena Shah, Professor, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT2016MS2
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Condition (Experimental)
  Interventions: Other: Exercise Condition
- Control Condition (Active Comparator)
  Interventions: Other: Control Condition

INTERVENTIONS:
Other: Exercise Condition — A bout of exercise in the evening followed by high-sugar meal consumption the following morning
  Arms: Exercise Condition
Other: Control Condition — Rest in the evening followed by high-sugar meal consumption the following morning
  Arms: Control Condition

SUMMARY:
The purpose of this study is to determine if postprandial (after a meal) endothelial (inner lining of blood vessels) dysfunction induced by a high sugar meal improves with a bout of exercise

DETAILED DESCRIPTION:
Endothelial dysfunction is due to an imbalance between vasodilating and vasoconstricting substances produced by the endothelium. An imbalance in these substances limits the ability of the blood vessel to relax in response to a shear stress stimulus. Endothelial dysfunction is a major risk factor for cardiovascular disease.

High-sugar intakes result in postprandial hyperglycemia and endothelial dysfunction. Exercise may attenuate the endothelial dysfunction induced by a high-sugar meal. There are only two studies that have examined the effect of exercise on endothelial dysfunction induced by high-sugar intake. Both studies found that a bout of aerobic exercise attenuated the impaired flow mediated dilation induced by high-sugar ingestion. Neither study measured important markers of endothelial dysfunction such as blood nitric oxide, endothelin I, and angiotensin II concentrations, however. In addition, whether the same results apply to older post-menopausal women is unknown. Understanding how acute exercise affects meal-induced endothelial dysfunction in older women is important given that age is related to endothelial dysfunction and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* Must be 45-70 years

Exclusion Criteria:

* Use of medications or supplements to lose weight
* Following a weight loss diet
* Smoking
* Heavy alcohol consumption
* Diabetes
* Heart disease
* Stroke
* Liver disease
* Kidney disease
* Untreated thyroid disease
* Anemia
* Uncontrolled hypertension
* Pulmonary disease that prevents exercise
* Orthopedic problems that prevents exercise
* Arthritis problems that prevent exercise
* Musculoskeletal problems that prevent exercise.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery flow mediated dilation | 0, 60, 120, and 180 minutes

SECONDARY OUTCOMES:
Change in blood nitric oxide concentration | 0, 60, 120, and 180 minutes
Change in blood endothelin-1concentration | 0, 60, 120, and 180 minutes
Change in blood angiotensin II concentration | 0, 60, 120, and 180 minutes
Change in blood glucose concentration | 0, 60, 120, and 180 minutes
Change in blood insulin concentration | 0, 60, 120, and 180 minutes
Change in blood lipoprotein particle numbers | 0, 60, 120, and 180 minutes
Change in blood lipid concentration | 0, 60, 120, and 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Meena Shah, Ph.D., Principal Investigator — Tzu Chi University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

REFERENCES:
- [Background] Deanfield J, Donald A, Ferri C, Giannattasio C, Halcox J, Halligan S, Lerman A, Mancia G, Oliver JJ, Pessina AC, Rizzoni D, Rossi GP, Salvetti A, Schiffrin EL, Taddei S, Webb DJ; Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. Endothelial function and dysfunction. Part I: Methodological issues for assessment in the different vascular beds: a statement by the Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. J Hypertens. 2005 Jan;23(1):7-17. doi: 10.1097/00004872-200501000-00004. PMID 15643116
- [Background] Widmer RJ, Lerman A. Endothelial dysfunction and cardiovascular disease. Glob Cardiol Sci Pract. 2014 Oct 16;2014(3):291-308. doi: 10.5339/gcsp.2014.43. eCollection 2014. No abstract available. PMID 25780786
- [Background] Loader J, Montero D, Lorenzen C, Watts R, Meziat C, Reboul C, Stewart S, Walther G. Acute Hyperglycemia Impairs Vascular Function in Healthy and Cardiometabolic Diseased Subjects: Systematic Review and Meta-Analysis. Arterioscler Thromb Vasc Biol. 2015 Sep;35(9):2060-72. doi: 10.1161/ATVBAHA.115.305530. Epub 2015 Jun 25. PMID 26112007
- [Background] Zhu W, Zhong C, Yu Y, Li K. Acute effects of hyperglycaemia with and without exercise on endothelial function in healthy young men. Eur J Appl Physiol. 2007 Apr;99(6):585-91. doi: 10.1007/s00421-006-0378-3. Epub 2007 Jan 6. PMID 17206439
- [Background] Weiss EP, Arif H, Villareal DT, Marzetti E, Holloszy JO. Endothelial function after high-sugar-food ingestion improves with endurance exercise performed on the previous day. Am J Clin Nutr. 2008 Jul;88(1):51-7. doi: 10.1093/ajcn/88.1.51. PMID 18614723
- [Derived] Shah M, Gloeckner A, Bailey S, Adams-Huet B, Kreutzer A, Cheek D, Willis JL, Mitchell J. Effect of a late afternoon/early evening bout of aerobic exercise on postprandial lipid and lipoprotein particle responses to a high-sugar meal breakfast the following day in postmenopausal women: a randomized cross-over study. J Sports Sci. 2022 Jan;40(2):175-184. doi: 10.1080/02640414.2021.1982497. Epub 2021 Sep 27. PMID 34565292
- [Derived] Shah M, Bailey S, Gloeckner A, Kreutzer A, Adams-Huet B, Cheek D, Mitchell J. Effect of acute exercise on postprandial endothelial function in postmenopausal women: a randomized cross-over study. J Investig Med. 2019 Aug;67(6):964-970. doi: 10.1136/jim-2019-000992. Epub 2019 Mar 5. PMID 30842213